CLINICAL TRIAL: NCT04617080
Title: Prospective Clinical Study to Evaluate the Safety and Efficacy of Different Add Powers With a New Presbyopic Lasik Treatment Algorithm
Brief Title: Safety and Efficacy of Different Add Powers With a New Presbyopic Lasik Treatment Algorithm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL1901
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUPRACOR Regular (Active Comparator)
  Interventions: Procedure: SUPRACOR Regular
- SUPRACOR Strong (Experimental)
  Interventions: Procedure: SUPRACOR Strong

INTERVENTIONS:
Procedure: SUPRACOR Regular — SUPRACOR algorithm with regular (100%) ablation profile. SUPRACOR is a presbyopic algorithm that consists of a pre-calculated pulse pattern combined to the refractive pattern to combine near, intermediate and distance vision correction.
  Arms: SUPRACOR Regular
Procedure: SUPRACOR Strong — SUPRACOR algorithm with strong (130%) ablation profile. SUPRACOR is a presbyopic algorithm that consists of a pre-calculated pulse pattern combined to the refractive pattern to combine near, intermediate and distance vision correction.
  Arms: SUPRACOR Strong

SUMMARY:
This is a prospective, comparative, randomized, controlled, open-label, single-surgeon, single-center PMCF clinical study whereby presbyopic patients undergoing refractive surgery will receive a SUPRACOR treatment for the correction in the non-dominant eye and a PROSCAN refractive treatment in the dominant eye to correct for ametropia.

The participants will be randomized to either a SUPRACOR regular (100%) or SUPRACOR strong (130%) treatment with a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* presbyopia
* willingness for a refractive presbyopia correction
* signed informed consent form

Exclusion Criteria:

- ocular comorbidity

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-26 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Binocular Uncorrected Distance Visual Acuity (UDVA) | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under photopic light conditions.

SECONDARY OUTCOMES:
Monocular Uncorrected Distance Visual Acuity (UDVA) | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under photopic light conditions.
Monocular Corrected Distance Visual Acuity (CDVA) | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under photopic light conditions. Corrected means spectacle corrected.
Binocular Corrected Distance Visual Acuity (CDVA) | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under photopic light conditions. Corrected means spectacle corrected.
Monocular Uncorrected Intermediate Visual Acuity (UIVA) | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 80 cm (intermediate distance) in LogMAR scale under photopic light conditions.
Binocular Uncorrected Intermediate Visual Acuity (UIVA) | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 80 cm (intermediate distance) in LogMAR scale under photopic light conditions.
Monocular Uncorrected Near Visual Acuity (UNVA) | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 40 cm (near distance) in LogMAR scale under photopic light conditions.
Binocular Uncorrected Near Visual Acuity (UNVA) | 3 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 40 cm (near distance) in LogMAR scale under photopic light conditions.
Binocular Defocus Curve | 3 months follow up
  To assess the visual acuity for different distances, defocus curves under photopic light conditions will be measured using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) device at 4m. This test is performed with best distance corrected refraction and spherical additions ranging from -4.5 D to +1.0 D in 0.5D steps.
Binocular Contrast sensitivity | 3 months follow up
  The contrast sensitivity test consists in assessing the possibility to distinguish the alternation of white and grey fringes of difference contrast with difference frequency. Contrast sensitivity will be assessed under photopic and mesopic light conditions using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) device at 2.5 m.
Halo Photic phenomena | 3 months follow up
  The amount and disturbance of photic halo side effects will be assessed by two methods: 1) Halo and Glare simulator: With this software tool the particant mimics the individual vision perception by adjusting a typical night scene image with the intensity and size of glare and halo; 2) Siepser Glarometer (Gulden Ophthalmics, Elkins Park, PA 19027). This is a target-like device that measures and quantifies post-operative glare. The measurement is of the participants' actual scope and range of monocular glare and halo.
Glare Photic phenomena | 3 months follow up
  The amount and disturbance of photic glare side effects will be assessed by two methods: 1) Halo and Glare simulator: With this software tool the particant mimics the individual vision perception by adjusting a typical night scene image with the intensity and size of glare and halo; 2) Siepser Glarometer (Gulden Ophthalmics, Elkins Park, PA 19027). This is a target-like device that measures and quantifies post-operative glare. The measurement is of the participants' actual scope and range of monocular glare and halo.
Patient-Reported Spectacle Independence Questionnaire (PRSIQ) | 3 months follow up
  The Patient-Reported Spectacle Independence Questionnaire (PRSIQ) is comprised of 3 questions about the need for glasses or contacts in the past 7 days for distance vision (at least 1.5 meters (m) away), intermediate vision (0.5 m to 1.5 m away), and near vision (< 0.5 m away). Possible scores range from 1 to 5, with 1 = All of the time and 5 = None of the time for six of the questions; 3 of these questions ask the question in a positive way and 3 of the question ask the question in a negative way, so the higher scores are better for the negative question and are worse for the positive question. There are also 3 questions whether glasses or contacts were needed in the past 7 days with scores of Yes = 1 and No = 2. The results for each question will be summarized separately.
Near Activity Visual Questionnaire (NAVQ) | 3 months follow up
  The Near Activity Visual Questionnaire (NAVQ) is comprised of 10 questions about performing activities without extra reading spectacles. Each question has responses of 0 to 4, with 0 indicating 'No difficulty' and 4 indicating 'Extreme difficulty'. Any 'Not applicable' responses are scored according to the median overall score for the subject. The scores are summed with total score ranging from 0 to 30. Higher scores indicate more difficulty performing specified activities without spectacles.

OTHER OUTCOMES:
Binocular Uncorrected Distance Visual Acuity (UDVA) | 12 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under photopic light conditions.
Monocular Uncorrected Distance Visual Acuity (UDVA) | 12 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m in LogMAR scale under photopic light conditions.
Monocular Corrected Distance Visual Acuity (CDVA) | 12 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m, 80 cm and 40 cm in LogMAR scale under photopic light conditions. Corrected means spectacle corrected.
Binocular Corrected Distance Visual Acuity (CDVA) | 12 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 4 m, 80 cm and 40 cm in LogMAR scale under photopic light conditions. Corrected means spectacle corrected.
Monocular Uncorrected Intermediate Visual Acuity (UIVA) | 12 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 80 cm (intermediate distance) in LogMAR scale under photopic light conditions.
Binocular Uncorrected Intermediate Visual Acuity (UIVA) | 12 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 80 cm (intermediate distance) in LogMAR scale under photopic light conditions.
Monocular Uncorrected Near Visual Acuity (UNVA) | 12 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 40 cm (near distance) in LogMAR scale under photopic light conditions.
Binocular Uncorrected Near Visual Acuity (UNVA) | 12 months follow up
  The visual acuity measurements will be assessed using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) at 40 cm (near distance) in LogMAR scale under photopic light conditions.
Binocular Defocus Curve | 12 months follow up
  To assess the visual acuity for different distances, defocus curves under photopic light conditions will be measured using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) device at 4m. This test is performed with best distance corrected refraction and spherical additions ranging from -4.5 D to +1.0 D in 0.5D steps.
Binocular Contrast sensitivity | 12 months follow up
  The contrast sensitivity test consists in assessing the possibility to distinguish the alternation of white and grey fringes of difference contrast with difference frequency. Contrast sensitivity will be assessed under photopic and mesopic light conditions using Clinical Trial Suite (M&S Technologies, Niles, IL, USA) device at 2.5 m.
Halo Photic phenomena | 12 months follow up
  The amount and disturbance of photic halo side effects will be assessed by two methods: 1) Halo and Glare simulator: With this software tool the particant mimics the individual vision perception by adjusting a typical night scene image with the intensity and size of glare and halo; 2) Siepser Glarometer (Gulden Ophthalmics, Elkins Park, PA 19027). This is a target-like device that measures and quantifies post-operative glare. The measurement is of the participants' actual scope and range of monocular glare and halo.
Glare Photic phenomena | 12 months follow up
  The amount and disturbance of photic glare side effects will be assessed by two methods: 1) Halo and Glare simulator: With this software tool the particant mimics the individual vision perception by adjusting a typical night scene image with the intensity and size of glare and halo; 2) Siepser Glarometer (Gulden Ophthalmics, Elkins Park, PA 19027). This is a target-like device that measures and quantifies post-operative glare. The measurement is of the participants' actual scope and range of monocular glare and halo.
Patient-Reported Spectacle Independence Questionnaire (PRSIQ) | 12 months follow up
  The Patient-Reported Spectacle Independence Questionnaire (PRSIQ) is comprised of 3 questions about the need for glasses or contacts in the past 7 days for distance vision (at least 1.5 meters (m) away), intermediate vision (0.5 m to 1.5 m away), and near vision (< 0.5 m away). Possible scores range from 1 to 5, with 1 = All of the time and 5 = None of the time for six of the questions; 3 of these questions ask the question in a positive way and 3 of the question ask the question in a negative way, so the higher scores are better for the negative question and are worse for the positive question. There are also 3 questions whether glasses or contacts were needed in the past 7 days with scores of Yes = 1 and No = 2. The results for each question will be summarized separately.
Near Activity Visual Questionnaire (NAVQ) | 12 months follow up
  The Near Activity Visual Questionnaire (NAVQ) is comprised of 10 questions about performing activities without extra reading spectacles. Each question has responses of 0 to 4, with 0 indicating 'No difficulty' and 4 indicating 'Extreme difficulty'. Any 'Not applicable' responses are scored according to the median overall score for the subject. The scores are summed with total score ranging from 0 to 30. Higher scores indicate more difficulty performing specified activities without spectacles.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ang, MD, Principal Investigator — Asian Eye Institute
Locations (1):
- Asian Eye Institute, Makati City, Philippines

IPD SHARING:
Plan to Share IPD: Undecided